CLINICAL TRIAL: NCT03478787
Title: A Multicenter, Randomized, Open Label, Efficacy Assessor-Blinded Study of Risankizumab Compared to Secukinumab for the Treatment of Adult Subjects With Moderate to Severe Plaque Psoriasis Who Are Candidates for Systemic Therapy
Brief Title: Risankizumab Versus Secukinumab for Participants With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M16-766; 2017-004932-12 (EudraCT Number)
Record Dates: First submitted 2018-03-23; First posted 2018-03-27 (Actual); Results first posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-06

CONDITIONS: Psoriasis
Keywords: Plaque Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — risankizumab; secukinumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Risankizumab (Experimental): Participants randomized to risankizumab receive 2 injections of active risankizumab (150 mg total dosage) subcutaneously (SC) at Weeks 0 and 4, and then every 12 weeks (q12w) thereafter until the last dose at Week 40 (Week 64 for participants in France).
  Interventions: Drug: risankizumab
- Secukinumab (Active Comparator): Participants randomized to secukinumab receive 2 injections of active secukinumab (300 mg total dosage) SC at Weeks 0, 1, 2, 3, and 4, and then every 4 weeks (q4w) thereafter until the last dose at Week 48.
  Interventions: Drug: secukinumab

INTERVENTIONS:
Drug: risankizumab — Subcutaneous (SC) injection
  Other Names: ABBV-066; BI 655066; SKYRIZI
  Arms: Risankizumab
Drug: secukinumab — Subcutaneous (SC) injection
  Other Names: Cosentyx
  Arms: Secukinumab

SUMMARY:
The main objective of this study is to evaluate the efficacy and safety of risankizumab compared with secukinumab for the treatment of adult subjects with moderate to severe plaque psoriasis who are candidates for systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic plaque psoriasis with or without psoriatic arthritis for at least 6 months before the Baseline Visit
* Subject has stable moderate to severe chronic plaque psoriasis with or without psoriatic arthritis
* Subject must be a candidate for systemic therapy as assessed by the investigator;
* Subject must be an acceptable candidate to receive secukinumab according to the local label for this compound.

Exclusion Criteria:

* History of erythrodermic psoriasis, generalized or localized pustular psoriasis, medication-induced or medication-exacerbated psoriasis, or new onset guttate psoriasis; or active skin disease other than psoriasis that could interfere with the assessment of psoriasis;
* Chronic infections including HIV, viral hepatitis (hepatitis B, hepatitis C), and/ or active tuberculosis. Subjects with a positive QuantiFERON®-TB/purified protein derivative (PPD) test result may participate in the study if further work up (according to local practice/guidelines) establishes conclusively that the subject has no evidence of active tuberculosis. If presence of latent tuberculosis is established, then treatment must have been initiated and maintained according to local country guidelines.
* Active systemic infection during the last 2 weeks prior to Baseline Visit (exception: common cold)
* History of any documented active or suspected malignancy or history of any malignancy within the last 5 years except for successfully treated non-melanoma skin cancer (NMSC) or localized carcinoma in situ of the cervix
* Previous exposure to risankizumab
* Previous exposure to secukinumab

Min Age: 18 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2020-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (61):
- United States (28):
  - Advanced Research Associates - Glendale /ID# 204335, Glendale, Arizona
  - Alliance Dermatology and MOHs /ID# 204336, Phoenix, Arizona
  - Bakersfield Derma & Skin Cance /ID# 202115, Bakersfield, California
  - Center for Dermatology Clin Res /ID# 202116, Fremont, California
  - Dermatology Res. Assoc., CA /ID# 202170, Los Angeles, California
  - UC Davis Health /ID# 202263, Sacramento, California
  - Medderm Associates /ID# 202162, San Diego, California
  - UConn Health Main /ID# 201745, Farmington, Connecticut
  - Tory P Sullivan, MD PA /ID# 202177, North Miami Beach, Florida
  - Renstar Medical Research /ID# 202113, Ocala, Florida
  - Progressive Medical Research /ID# 202183, Port Orange, Florida
  - Integrated Clinical Research LLC /ID# 202152, West Palm Beach, Florida
  - Dermatology Specialists Resear /ID# 202145, Louisville, Kentucky
  - Dermatology and Skin Cancer Specialists, LLC /ID# 203938, Rockville, Maryland
  - ORA, Inc. /ID# 204342, Andover, Massachusetts
  - Beth Israel Deaconess Medical Center /ID# 204340, Boston, Massachusetts
  - Minnesota Clinical Study Center /ID# 202369, New Brighton, Minnesota
  - Central Dermatology, PC /ID# 202156, St Louis, Missouri
  - Psoriasis Treatment Ctr of Central NJ /ID# 202107, East Windsor, New Jersey
  - Synexus Research Cincinnati /ID# 202161, Cincinnati, Ohio
  - Oregon Derm & Res. Ctr /ID# 201652, Portland, Oregon
  - Oregon Medical Res Center PC /ID# 201651, Portland, Oregon
  - Clinical Partners, LLC /ID# 201736, Johnston, Rhode Island
  - Center for Clinical Studies - Houston (Binz) /ID# 202178, Houston, Texas
  - Progressive Clinical Research /ID# 202155, San Antonio, Texas
  - Center for Clinical Studies - Webster TX /ID# 202154, Webster, Texas
  - University of Utah /ID# 204035, Salt Lake City, Utah
  - Froedtert Mem Lutheran Hosp /ID# 204896, Milwaukee, Wisconsin
- Canada (7):
  - Beacon Dermatology Inc /ID# 203054, Calgary, Alberta
  - Enverus Medical Research /ID# 203043, Surrey, British Columbia
  - Dr. Irina Turchin PC Inc. /ID# 203052, Fredericton, New Brunswick
  - Eastern Canada Cutaneous Resea /ID# 203045, Halifax, Nova Scotia
  - Dermatrials Research /ID# 203051, Hamilton, Ontario
  - Dre Angelique Gagne-Henley M.D. inc. /ID# 203053, Saint-Jérôme, Quebec
  - Dermatologique du Quebec /ID# 203050, Québec
- France (5):
  - Charles Nicolle CHU Rouen /ID# 203590, Rouen, Seine-Maritime
  - Centre Hospitalier Universitaire de Nice - Hopital l'Archet 2 /ID# 203591, Nice
  - Hopital Saint-Louis /ID# 203586, Paris
  - Polyclinique Courlancy /ID# 203588, Reims
  - Hopital Larrey - CHU de Toulouse /ID# 203587, Toulouse
- TU Uniklinik Munchen /ID# 203919, Munich, Germany
- Italy (2):
  - Policlinico A. Gemelli /ID# 203009, Rome, Lazio
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico /ID# 204982, Milan, Lombardy
- Netherlands (3):
  - Radboud Universitair Medisch Centrum /ID# 202560, Nijmegen, Gelderland
  - Bravis Ziekenhuis /ID# 205232, Bergen op Zoom, North Brabant
  - Academisch Medical center Amsterdam /ID# 202556, Amsterdam, North Holland
- Poland (6):
  - Klinika Dermatologii Pod Fortem /ID# 204180, Krakow, Lesser Poland Voivodeship
  - Przychodnia Specjalistyczna High-Med /ID# 203183, Warsaw, Masovian Voivodeship
  - Klinika Ambroziak Sp. z o.o. /ID# 203928, Warsaw, Masovian Voivodeship
  - KSW nr1 w Rzeszowie /ID# 203776, Rzeszów, Podkarpackie Voivodeship
  - Osteo-Medic S.C. /ID# 203742, Bialystok, Podlaskie Voivodeship
  - Dermed Centrum Medyczne Sp. z o.o /ID# 203171, Lodz, Łódź Voivodeship
- Spain (6):
  - Hospital de Manises /ID# 203757, Manises, Valencia
  - Hospital General Universitario Alicante /ID# 203764, Alicante
  - Hospital Universitario Clinico San Cecilio /ID# 203760, Granada
  - Hospital Universitario de la Princesa /ID# 203754, Madrid
  - Hospital Universitario 12 de Octubre /ID# 203756, Madrid
  - Hospital Universitario Arnau Vilanova /ID# 203763, Valencia
- United Kingdom (3):
  - Whipps Cross Univ Hospital /ID# 204723, London, London, City of
  - Guy's and St Thomas' NHS Found /ID# 204721, London, London, City of
  - The University of Manchester /ID# 204720, Salford

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Crowley JJ, Langley RG, Gordon KB, Pinter A, Ferris LK, Rubant S, Photowala H, Xue Z, Wu T, Zhan T, Beeck S, Shah M, Warren RB. Efficacy of Risankizumab versus Secukinumab in Patients with Moderate-to-Severe Psoriasis: Subgroup Analysis from the IMMerge Study. Dermatol Ther (Heidelb). 2022 Feb;12(2):561-575. doi: 10.1007/s13555-021-00679-6. Epub 2022 Jan 20. PMID 35050485

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 327 participants were randomized from 53 sites across 9 countries including Canada, France, Germany, Italy, The Netherlands, Poland, Spain, the United Kingdom, and the United States.
Pre-assignment Details: Eligible participants were randomized to receive risankizumab or secukinumab in a 1:1 ratio. The randomization was stratified by weight (≤ 100 kg vs. > 100 kg) and prior systemic biologic for psoriasis (0 vs. ≥ 1).
Groups:
- Secukinumab: Participants randomized to secukinumab received 2 injections of active secukinumab (300 mg total dosage) subcutaneously (SC) at Weeks 0, 1, 2, 3, and 4, and then every 4 weeks (q4w) thereafter until the last dose at Week 48.
- Risankizumab: Participants randomized to risankizumab received 2 injections of active risankizumab (150 mg total dosage) SC at Weeks 0 and 4, and then every 12 weeks (q12w) thereafter until the last dose at Week 40 (Week 64 for participants in France).
Period: Overall Study
Arm/Group | Secukinumab | Risankizumab
Started | 163 | 164
Completed | 134 | 151
Not Completed | 29 | 13
Not completed — Adverse Event | 5 | 1
Not completed — Protocol Violation | 3 | 0
Not completed — Lack of Efficacy | 7 | 1
Not completed — Lost to Follow-up | 9 | 5
Not completed — Withdrawal by Subject | 2 | 6
Not completed — Other, Not Specified | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab | Risankizumab | Total
Number analyzed (Participants) | 163 | 164 | 327
Age, Customized [Count of Participants; unit: Participants]
  < 40 years | 60 | 50 | 110
  40 to < 65 years | 81 | 99 | 180
  >/= 65 years | 22 | 15 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 52 | 114
  Male | 101 | 112 | 213
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 37 | 71
  Not Hispanic or Latino | 129 | 127 | 256
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 11 | 6 | 17
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 6 | 6 | 12
  White | 144 | 151 | 295
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a 90% Reduction From Baseline Psoriasis Area and Severity Index (PASI 90) at Week 16
Description: The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI 90 is defined as at least a 90% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100. Non-responder imputation (NRI) was used for missing data.
Time Frame: Week 16
Population: Intent to Treat (ITT) analysis set: all participants who were randomized at Baseline. Non-responder imputation (NRI) was used for missing data.
Measure: Number; unit: percentage of participants
Arm/Group | Secukinumab | Risankizumab
Number analyzed (Participants) | 163 | 164
percentage of participants | 65.6 | 73.8
Statistical Analysis 1: Comparison: Secukinumab vs Risankizumab; Test type: Non-Inferiority — Non-inferiority is met if the lower bound of the 96.25% confidence interval (CI) of adjusted treatment difference is above -12%; Adjusted percentage difference = 8.2, 96.25% CI 2-sided [-2.2 to 18.6] — Across the strata, 96.25% confidence interval (CI) for adjusted difference was calculated according to the Cochran-Mantel-Haenszel test for the comparison of 2 treatment groups

2. Primary Outcome: Percentage of Participants With a PASI 90 at Week 52
Description: The PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI 90 is defined as at least a 90% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100.
Time Frame: Week 52
Population: ITT analysis set: all participants who were randomized at Baseline. NRI was used for missing data.
Measure: Number; unit: percentage of participants
Arm/Group | Secukinumab | Risankizumab
Number analyzed (Participants) | 163 | 164
percentage of participants | 57.1 | 86.6
Statistical Analysis 1: Comparison: Secukinumab vs Risankizumab; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Across the strata, p-value was calculated from the from the Cochran-Mantel-Haenszel test adjusted for strata; Adjusted percentage difference = 29.8, 95% CI 2-sided [20.8 to 38.8] — Across the strata, 95% CI for adjusted difference was calculated according to the Cochran-Mantel-Haenszel test for the comparison of 2 treatment groups

3. Secondary Outcome: Percentage of Participants With a 100% Reduction From Baseline Psoriasis Area and Severity Index (PASI 100) at Week 52
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI 100 is defined as 100% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100.
Time Frame: Week 52
Population: ITT analysis set: all participants who were randomized at Baseline. NRI was used for missing data.
Measure: Number; unit: percentage of participants
Arm/Group | Secukinumab | Risankizumab
Number analyzed (Participants) | 163 | 164
percentage of participants | 39.9 | 65.9
Statistical Analysis 1: Comparison: Secukinumab vs Risankizumab; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Across the strata, p-value was calculated from the from the Cochran-Mantel-Haenszel test adjusted for strata; Adjusted percentage difference = 26.2, 95% CI 2-sided [15.9 to 36.5] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Percentage of Participants Achieving Static Physician Global Assessment (sPGA) of Clear or Almost Clear at Week 52
Description: The sPGA is an assessment by the investigator of the overall disease severity at the time of evaluation. Erythema, induration, and scaling of psoriatic lesions are scored on a 5-point scale ranging from 0 (none) to 4 (severe). The sPGA ranges from 0 to 4, and is calculated as Clear (0) = 0 for all 3; Almost clear (1) = mean > 0, < 1.5; Mild (2) = mean ≥ 1.5, < 2.5; Moderate (3) = mean ≥ 2.5, < 3.5; and Severe (4) = mean ≥ 3.5.
Time Frame: Week 52
Population: ITT analysis set: all participants who were randomized at Baseline. NRI was used for missing data.
Measure: Number; unit: percentage of participants
Arm/Group | Secukinumab | Risankizumab
Number analyzed (Participants) | 163 | 164
percentage of participants | 58.3 | 87.8
Statistical Analysis 1: Comparison: Secukinumab vs Risankizumab; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Across the strata, p-value was calculated from the from the Cochran-Mantel-Haenszel test adjusted for strata; Adjusted percentage difference = 29.8, 95% CI 2-sided [20.9 to 38.8] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Percentage of Participants With a 75% Reduction From Baseline Psoriasis Area and Severity Index (PASI 75) at Week 52
Description: The PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI 75 is defined as at least a 75% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100.
Time Frame: Week 52
Population: ITT analysis set: all participants who were randomized at Baseline. NRI was used for missing data.
Measure: Number; unit: percentage of participants
Arm/Group | Secukinumab | Risankizumab
Number analyzed (Participants) | 163 | 164
percentage of participants | 69.9 | 89.6
Statistical Analysis 1: Comparison: Secukinumab vs Risankizumab; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Across the strata, p-value was calculated from the from the Cochran-Mantel-Haenszel test adjusted for strata; Adjusted percentage difference = 20.0, 95% CI 2-sided [11.7 to 28.3] — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are reported from first dose of study drug through 20 weeks after last dose of study drug (up to Week 68 for the Secukinumab arm, and up to Week 84 for the Risankizumab arm).
Groups:
- Secukinumab: Participants randomized to secukinumab received 2 injections of active secukinumab (300 mg total dosage) subcutaneously (SC) at Weeks 0, 1, 2, 3, and 4, and then every 4 weeks (q4w) thereafter until the last dose at Week 48 and received at least one dose of study drug.
- Risankizumab: Participants randomized to risankizumab received 2 injections of active risankizumab (150 mg total dosage) SC at Weeks 0 and 4, and then every 12 weeks (q12w) thereafter until the last dose at Week 40 (Week 64 for participants in France) and received at least one dose of study drug .
Arm/Group | Secukinumab | Risankizumab
All-Cause Mortality (participants affected / at risk) | 0/163 | 0/164
Serious Adverse Events (participants affected / at risk) | 6/163 | 9/164
Other Adverse Events (participants affected / at risk) | 71/163 | 66/164
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Secukinumab (N=163) | Risankizumab (N=164)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1)
ARRHYTHMIA SUPRAVENTRICULAR (Cardiac disorders) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1)
BASEDOW'S DISEASE (Endocrine disorders) | 0 (0) | 1 (1)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIVERTICULUM INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 1 (1) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 2 (2)
OVERDOSE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HISTIOCYTIC NECROTISING LYMPHADENITIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
TOXIC ENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 0 (0)
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 (0) | 1 (1)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 1 (1)
SUICIDE ATTEMPT (Psychiatric disorders) | 0 (0) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1)
OVARIAN CYST (Reproductive system and breast disorders) | 0 (0) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ARTERIOSCLEROSIS (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Secukinumab (N=163) | Risankizumab (N=164)
DIARRHOEA (Gastrointestinal disorders) | 9 (12) | 9 (11)
BRONCHITIS (Infections and infestations) | 11 (11) | 3 (3)
NASOPHARYNGITIS (Infections and infestations) | 27 (38) | 35 (48)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 14 (20) | 21 (25)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 10 (13) | 9 (12)
HEADACHE (Nervous system disorders) | 15 (27) | 9 (20)
HYPERTENSION (Vascular disorders) | 5 (5) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2019-08-16): https://cdn.clinicaltrials.gov/large-docs/87/NCT03478787/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-22): https://cdn.clinicaltrials.gov/large-docs/87/NCT03478787/SAP_001.pdf